CLINICAL TRIAL: NCT05373368
Title: How Quality of Life of Elderly Individuals Living at Home or in Nursing Homes is Related to Multi Purpose Activities?
Brief Title: Quality of Life Related to Activities of Elderly Individuals Living at Home or Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hulya Yucel, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07.T09.102.001
Record Dates: First submitted 2022-05-08; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Elderly; Quality of Life; Physical Activity
Keywords: Elderly; Leisure activity; Quality of life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home residents (Experimental): multi purpose activities were performed for home residents
  Interventions: Behavioral: multi purpose activities
- nursing home residents (Experimental): multi purpose activities were performed for nursing home residents
  Interventions: Behavioral: multi purpose activities

INTERVENTIONS:
Behavioral: multi purpose activities

SUMMARY:
For older persons, successful aging generally involves staying active and maintaining social interactions. Active aging involves more engagement in enjoyable activities. The hypothesis of this study was to determine the effects of multi-purpose activities on the quality of life of elderly individuals living either in a nursing home or in their own homes. Sixty-seven volunteers aged >60 were surveyed: 34 living in a nursing home and 33 living at-home. Participants performed activities consisting of physical, cognitive tasks, and handicrafts twice weekly for 12 weeks. Each participant completed the 36-item Short Form Health Survey both before and after the program, and the results were compared between the groups.

DETAILED DESCRIPTION:
In this study, investigators performed multi-purpose activity programs to see the effects on the quality of life (QOL) of the older persons. Eighty-one participants aged >60 residing in Ankara volunteered to participate in: 45 at the a nursing home, and 36 living in their own homes in the town. The investigators received participants' information from their files or from relatives to verify their eligibility criteria for this randomized study. The ethical review committee of Hacettepe University approved the study and written informed consent was obtained from each participant. This study was performed in accordance with the Declaration of Helsinki.

The collected socio-demographic data included age, gender, co-morbidities, years of schooling completed, and marital status. The 36-item Short Form Health Survey (SF 36) was used prior to and following the program in order to evaluate participants' QOL. Its eight parameters cover general health, physical functioning, vitality, physical role, physical energy level, social functioning, emotional role, and mental health. Higher scores indicate better functioning.

A therapist led the activity programs according to participants' requests and needs. Over twice-weekly 45-minute sessions for a period of 12 weeks, participants performed chosen activities in a group from the following three categories:

1. Handicrafts: ornament design, painting on cloth or glass, knitting, lace making, constructing book braces or vase base plates, arts, or woodwork.
2. Physical activities: gardening or dance.
3. Cognitive activities: puzzles (jigsaw and crossword), table games (backgammon and chess), watching classic movies, reading books, writing in diaries, or reminiscence activities.

The "General Health" sub-parameter of SF-36 was chosen to calculate the change between groups to determine the sample size, since this is theoretically the item with the widest range in mean and standard deviation. In the literature, the least level for measuring significant intra-group differences prior to and following a study intervention was 5 ± 8 points. With this information, investigators determined a sample size of 30 individuals per group was needed in order to have the correct power and confidence levels (90% and 95%, respectively) to detect a statistically significant difference using a 0.05 cut-off . Statistical analysis was performed using SPSS for Windows v. 23. Descriptive data were presented as mean (X) ± standard deviation (SD). Categorical data were presented as counts and percentages. The independent t-test was used to compare the QOL of at-home residents with those in the nursing home, and the Mann-Whitney U test was used if the parametric test assumptions are not ensured. A dependent t-test was used to analyze results prior to and following the activities program, and the Wilcoxon test was used when the parametric test assumptions were not ensured. P values <0.05 were considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* aged over 60 years and above
* individuals without physical, mental, or sensory integration disabilities that might interfere with their performance in activities

Exclusion Criteria:

* being un-volunteered
* aged below 60 years
* having comorbidities that interfere with activities

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
improved quality of life caused by participation in activities | 45 minutes
  Changes on the prior scores of quality of life assessed by SF-36, of the elderly at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hulya Yucel, Assoc. Prof., Principal Investigator — Saglik Bilimleri University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Effects of Recreational Exercises on the Strength, Flexibility, and Balance of Old-old Elderly Individuals — https://pubmed.ncbi.nlm.nih.gov/25364118/
- See also: The effects of physical activity on anxiety, depression, and quality of life in elderly people living in the community — https://pubmed.ncbi.nlm.nih.gov/30994779/
- See also: A study of physical activity, frailty, and health related quality of life among community-dwelling older adults in Taiwan — https://pubmed.ncbi.nlm.nih.gov/32941303/
- See also: Effects of a group-based physical and cognitive intervention on social activity and quality of life for elderly people with dementia in a geriatric health service facility: a quasi-randomised controlled trial. — https://pubmed.ncbi.nlm.nih.gov/33140499/